CLINICAL TRIAL: NCT02721706
Title: Cost-effectiveness Study of the CIPA Screening Method for Patients With Nutritional Risk at Hospital Admission
Brief Title: Cost-effectiveness Study of the New Nutrition Screening Tool CIPA at Hospital Admission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of the Nuestra Señora de Candelaria (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, José Pablo Suárez Llanos, Ph.D, M.D., University Hospital of the Nuestra Señora de Candelaria
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PI14/01226
Record Dates: First submitted 2016-03-01; First posted 2016-03-29 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Malnutrition
Keywords: Nutrition assessment; inpatients; cost-benefit analysis; quality of life; body composition; mass screening
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CIPA screening tool (Experimental): Patients are evaluated by CIPA nutritional screening tool
  Interventions: Other: CIPA nutritional screening tool
- usual hospital clinical care (No Intervention): Patients are not subject of CIPA screening tool, and continue the usual hospital clinical care

INTERVENTIONS:
Other: CIPA nutritional screening tool — The new nutritional screening tool termed CIPA includes Control of food Intake, Protein, and Anthropometry (CIPA) results positive when at least one of the following parameters is met: control of food intake for 72 h <50%, serum albumin <3 g/dl, body mass index <18.5 kg/m2 or mid-upper arm circumference ≤ 22.5 cm.
  Arms: CIPA screening tool

SUMMARY:
Objectives: To evaluate the cost-effectiveness of implementing a malnutrition screening tool "CIPA" at the Hospital Universitario Nuestra Señora de la Candelaria (HUNSC), comparing the impact on health and the healthcare costs of hospitalised patients who are screened for malnutrition and of patients following standard clinical practice. Methodology: The study will consist of a controlled trial on patients admitted to the Internal Medicine and General and Digestive Surgery wards at the HUNSC. In both wards patients will be assigned to a control or to an intervention group. The control group will follow usual hospital clinical care, while the intervention group will be administered the screening tool "CIPA" for early detection of malnutrition cases and they will be treated according to the screening results. The following variables will be evaluated: length of stay in hospital, mortality, readmissions and in-hospital complications. Cost-effectiveness analysis will be undertaken measuring effectiveness by Quality-Adjusted Life Years (QALYs). Cost per patient will be measured by identifying health care resource utilisation, and the cost-effectiveness measure will be the Incremental Cost-Effectiveness Ratio (ICER). Investigators will calculate the incremental cost per QALY gained related to the intervention. This analysis will allow to quantify the costs (incurred and saved) related to the introduction of the malnutrition screening tool CIPA in the hospital context and to measure the health impact of screened patients.

ELIGIBILITY:
Inclusion Criteria:

* Formal consent to participate in the study.
* Patients admitted to the Internal Medicine or General Surgery wards.

Exclusion Criteria:

* Patients treated with nutritional support before CIPA screening is performed.
* Patients transferred from other wards.
* Patients with an expected length of stay less than 72 hours.
* CIPA screening unfeasible for any reason.
* Patients with poor short-term prognosis.
* Bed destination at hospital admission nonrandomized.
* Patients participating in other investigation study.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 823 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness measured by incremental Cost-effectiveness ratio (ICER) | up to 3 months after Hospital discharge time

SECONDARY OUTCOMES:
incidence of mortality | up to 3 months after Hospital discharge time
Quality of life measured by quality-adjusted life years (QALYs) | up to 3 months after Hospital discharge time
mean length of stay (days) | through study completion, an average of 13 days
incidence of readmissions | up to 3 months after hospital discharge time

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alvarez-Hernandez J, Planas Vila M, Leon-Sanz M, Garcia de Lorenzo A, Celaya-Perez S, Garcia-Lorda P, Araujo K, Sarto Guerri B; PREDyCES researchers. Prevalence and costs of malnutrition in hospitalized patients; the PREDyCES Study. Nutr Hosp. 2012 Jul-Aug;27(4):1049-59. doi: 10.3305/nh.2012.27.4.5986. PMID 23165541
- [Background] Suarez Llanos JP, Benitez Brito N, Oliva Garcia JG, Pereyra-Garcia Castro F, Lopez Frias MA, Garcia Hernandez A, Diaz Sirgo B, Llorente Gomez de Segura I. [Introducing a mixed nutritional screening tool (CIPA) in a tertiary hospital]. Nutr Hosp. 2014 May 1;29(5):1149-53. doi: 10.3305/nh.2014.29.5.7299. Spanish. PMID 24951997
- [Background] Benitez Brito N, Mora Mendoza A, Suarez Llanos JP, Delgado Brito I, Perez Mendez LI, Herrera Rodriguez EM, Oliva Garcia JG, Pereyra-Garcia Castro F. [CONCORDANCE IN THE RESULTS OF CONTROL INTAKE PERFORMANCE OF 72 H BY DIFFERENT HEALTH PROFESSIONALS IN A TERTIARY HOSPITAL]. Nutr Hosp. 2015 Dec 1;32(6):2893-7. doi: 10.3305/nh.2015.32.6.9740. Spanish. PMID 26667749
- [Background] van Bokhorst-de van der Schueren MA, Guaitoli PR, Jansma EP, de Vet HC. Nutrition screening tools: does one size fit all? A systematic review of screening tools for the hospital setting. Clin Nutr. 2014 Feb;33(1):39-58. doi: 10.1016/j.clnu.2013.04.008. Epub 2013 Apr 19. PMID 23688831
- [Background] Kruizenga HM, Seidell JC, de Vet HC, Wierdsma NJ, van Bokhorst-de van der Schueren MA. Development and validation of a hospital screening tool for malnutrition: the short nutritional assessment questionnaire (SNAQ). Clin Nutr. 2005 Feb;24(1):75-82. doi: 10.1016/j.clnu.2004.07.015. PMID 15681104
- [Background] Benitez Brito N, Suarez Llanos JP, Fuentes Ferrer M, Oliva Garcia JG, Delgado Brito I, Pereyra-Garcia Castro F, Caracena Castellanos N, Acevedo Rodriguez CX, Palacio Abizanda E. Relationship between Mid-Upper Arm Circumference and Body Mass Index in Inpatients. PLoS One. 2016 Aug 5;11(8):e0160480. doi: 10.1371/journal.pone.0160480. eCollection 2016. PMID 27494612
- [Derived] Suarez-Llanos JP, Benitez-Brito N, Vallejo-Torres L, Delgado-Brito I, Rosat-Rodrigo A, Hernandez-Carballo C, Ramallo-Farina Y, Pereyra-Garcia-Castro F, Carlos-Romero J, Felipe-Perez N, Garcia-Niebla J, Calderon-Ledezma EM, Gonzalez-Melian TJ, Llorente-Gomez de Segura I, Barrera-Gomez MA. Clinical and cost-effectiveness analysis of early detection of patients at nutrition risk during their hospital stay through the new screening method CIPA: a study protocol. BMC Health Serv Res. 2017 Apr 20;17(1):292. doi: 10.1186/s12913-017-2218-z. PMID 28424063